CLINICAL TRIAL: NCT00106054
Title: An Open-Label, Multi-Center Phase II Trial of Neoadjuvant Irinotecan in Combination With Infusional 5-FU, Leucovorin (Folfiri) Plus Bevacizumab in Patients With Unresectable Hepatic-Only Metastases of Colorectal Carcinoma
Brief Title: Neoadjuvant Colorectal Cancer With Unresectable Liver Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After 1 year only 2 subjects enrolled and treated thus no meaningful efficacy analyses could be performed.
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5961065
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Colorectal Neoplasms; Liver Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms | interventions — Fluorouracil; Leucovorin; Bevacizumab

INTERVENTIONS:
Drug: Combination therapy of irinotecan with 5-FU, leucovorin plus bevacizumab in the neoadjuvant setting.

SUMMARY:
The study was terminated early due to low enrollment with only 2 subjects enrolled and treated after being open for enrollment for over a year. Therefore, no meaningful efficacy analyses could be performed.

This trial is studying the effects (good and bad) of a combination of drugs, Irinotecan in combination with infusional 5-FU, leucovorin (FOLFIFI) plus Bevacizumab, for cancer of the colon or rectum that has spread to the liver only and is currently not able to be removed by surgery. All of the drugs that will be received in this research study have been approved in the United States for colorectal cancer, that has spread to other areas of the body, including the liver. Another reason for doing this study is to see if the chemotherapy drugs FOLFIFI plus Bevacizumab can sufficiently decrease the size of the cancer in the liver so that any tumor remaining can be completely removed with surgery and, if it can be removed whether doing so will prolong the time it takes the cancer to return and/or prolong the life of these patients. This trial is also looking at the genes of people who take part in this study, to see if it is possible to find out characteristics that can help predict whose cancer will respond well or not so well, and who will have more or less side effects to this chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1
* Histological documentation of adenocarcinoma of the colon or rectum. The primary site must have been confirmed to be in the large bowel

Exclusion Criteria:

* Prior systemic anticancer therapy for mCRC
* Prior hepatic surgery, chemoembolization, hepatic artery infusion, radiofrequency ablation or cryotherapy for liver metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To determine the rate of R0 resection or pathologically confirmed CR in patients with hepatic only metastases

SECONDARY OUTCOMES:
oTo determine the resectable rate, defined as the number of subjects with R0 resection, pathologically staged CR, or undergoing non-surgical ablative procedures with curative intent divided by the total number of evaluable subjects following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5961065&StudyName=Neoadjuvant+Colorectal+Cancer+with+Unresectable+Liver+Metastases%2E